CLINICAL TRIAL: NCT06640400
Title: A Clinical Study of the Efficacy of Cardiovascular Ultrasound Therapy on the Rehabilitation of Patients After PCI for Coronary Artery Disease
Brief Title: Cardiovascular Ultrasound for the Rehabilitation of Patients With Coronary Heart Disease After PCI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KYLL-202308-006
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Coronary Heart Disease
Keywords: cardiovascular ultrasound; PCI; rehabilitation; coronary heart disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group received cardiovascular ultrasound plus conventional drug therapy.
  Interventions: Device: Cardiovascular ultrasound
- Control group (No Intervention): The control group received conventional drug treatment.

INTERVENTIONS:
Device: Cardiovascular ultrasound — Participants in the intervention group will be treated with a medical LIPUS device (838C-M-L-I/II, Shenzhen, China) for 10 days in addition to conventional medical treatment. The ultrasound therapy instrument is equipped with a sound head comprising 5 transducer units, operating at an ultrasonic frequency of 0.84MHz with a sound intensity range of 1 W/cm2 -1.25 W/cm2. The therapeutic ultrasound sessions necessitate a controlled environmental temperature. Patients will assume the supine position, exposing the precordial region, with the five-pronged head positioned parallel to the heart&amp;#39;s long axis, covering the entire precordial region including the right and left coronary arterial trunks and the aortic root. The ultrasound therapy device operates in a pulsed mode, with each treatment session lasting 20 minutes, comprising 2 daily sessions for a total of 20 treatments.
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to learn the efficacy of cardiovascular ultrasound therapy on the rehabilitation of patients with coronary heart disease after PCI. It will also learn about the safety of cardiovascular ultrasound. The main questions it aims to answer are:

Whether cardiovascular ultrasound improves cardiac function and prognosis in patients with coronary artery disease after PCI? What medical problems will participants experience after using cardiovascular ultrasound therapy? Researchers will compare cardiovascular ultrasound to a placebo (sham stimulation) to see if cardiovascular ultrasound works to treat coronary artery disease after PCI.

Participants will:

Patients were treated with cardiovascular ultrasound or placebo from the 24th hour after PCI for 20 minutes twice a day for 10 days.

Examination and detection of serum inflammatory markers, endothelial function indicators, cardiac function, and heart rate variability at multiple time points (baseline (24 hours post-PCI), days 5 and 10 post-intervention, and months 1 and 3.

Their symptoms were recorded, and depression and anxiety were scored.

DETAILED DESCRIPTION:
Background Coronary heart disease (CHD) is one of the leading causes of mortality and disability and places a financial burden on the healthcare system. Although cardiovascular ultrasound has shown its effectiveness and safety in improving refractory angina, relevant clinical studies are rare, and clinical evidence is severely lacking.

Methods and design This is a prospective, parallel-group, randomized control trial. We will enroll 200 patients with coronary artery disease after PCI and randomize them into 2 groups. The intervention group was given usual practice combined with cardiovascular ultrasound intervention and the control group was given usual practice combined with empty stimulation intervention. We used hs-CRP and IL-6 levels in serum after 20 times treatments with LIPUS as the primary outcome measures. Serum myocardial injury indicators levels and blood lipids indicators levels, markers of endothelial function levels, inflammatory factor levels, hemodynamic Indicators, Echocardiogram, 6-minute walk test, Short-term Heart rate variability, and mental health assessment were secondary outcomes. The researchers tested the outcome indicators at baseline (24th hours after PCI), 5th and 10th days, and 1st and 3rd months after the intervention. Statistical analyses were performed using SPSS 26.0 statistical software.

Discussion This study is the first clinical study of the rehabilitation efficacy of cardiovascular ultrasound in the treatment of coronary heart disease after PCI. Given that the current clinical recovery mainly depends on the body's self-limiting and conventional symptomatic treatment, Cardiovascular ultrasound, as a new therapy method, might be a major advance in the treatment of coronary heart disease after PCI.

ELIGIBILITY:
Inclusion Criteria

1. Age of enrollment at least 18 years 2. Patients with confirmed coronary artery disease requiring elective PCI 3. TIMI flow grade 2 or above after PCI 4. No intraoperative complications of PCI such as entrapment, reflux, or perforation of coronary artery.

5. The skin in the anterior chest area is intact and not broken. 6. Cardiac enzymes and troponin I are within normal range before enrollment. Exclusion Criteria

1. Patients with ST-segment elevation myocardial infarction and non-ST-segment elevation myocardial infarction.
2. Occlusion of branch vessels during PCI.
3. Patients with perioperative use of hormones or immunosuppressants
4. Combined infection or other inflammatory diseases
5. Postoperative fever
6. Patients are allergic to contrast media or cardiovascular ultrasound acoustic head-related materials.
7. Changes in lipid-lowering, antiplatelet, and antihypertensive drug regimens during treatment.
8. Patients with a clear diagnosis of autoimmune disease
9. Patients who have undergone other surgeries in the past 7 days or have a history of trauma.
10. Patients infected with novel coronavirus in the past month.
11. Previous PCI treatment
12. Previous cardiovascular ultrasound treatment
13. Diabetic patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-25 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
high-sensitivity C-reactive protein (hs-CRP) in serum | Day 11 after PCI
  High-sensitivity C-reactive protein (hs-CRP) levels in serum following 20 cardiovascular ultrasound therapy treatment sessions.
Interleukin-6 (IL-6) levels | Day 11 after PCI
  high-sensitivity C-reactive protein (hs-CRP) and Interleukin-6 (IL-6) levels in serum following 20 cardiovascular ultrasound therapy treatment sessions

SECONDARY OUTCOMES:
creatine kinase isoenzymes | From enrollment to the end of treatment at 3rd month
  Serum creatine kinase isoenzyme levels in fasting were collected and measured
cardiac troponin I | From enrollment to the end of treatment at 3rd month
  Serum cardiac troponin I levels in fasting were collected and measured
myeloperoxidase | From enrollment to the end of treatment at 3rd month
  Serum myeloperoxidase levels in fasting were collected and measured.
total cholesterol | From enrollment to the end of treatment at 3rd month
  Serum total cholesterol levels in fasting were collected and measured
triglyceride | From enrollment to the end of treatment at 3rd month
  Serum triglyceride levels in fasting were collected and measured.
low-density lipoprotein cholesterol | From enrollment to the end of treatment at 3rd month
  Serum low-density lipoprotein cholesterol levels in fasting were collected and measured.
high-density lipoprotein cholesterol | From enrollment to the end of treatment at 3rd month
  Serum high-density lipoprotein cholesterol levels in fasting were collected and measured.
apolipoprotein A | From enrollment to the end of treatment at 3rd month
  Serum apolipoprotein A levels in fasting were collected and measured.
apolipoprotein B | From enrollment to the end of treatment at 3rd month
  Serum apolipoprotein B levels in fasting were collected and measured.
lipoprotein (a) | From enrollment to the end of treatment at 3rd month
  Serum lipoprotein (a) levels in fasting were collected and measured.
oxidized low-density lipoprotein | From enrollment to the end of treatment at 3rd month
  Serum-oxidized low-density lipoprotein levels in fasting were collected and measured.
endothelial nitric oxide synthase | From enrollment to the end of treatment at 3rd month
  Serum endothelial nitric oxide synthase levels in fasting were collected and measured.
endothelin-1 | From enrollment to the end of treatment at 3rd month
  Serum endothelin-1 levels in fasting were collected and measured.
vascular endothelial growth factor | From enrollment to the end of treatment at 3rd month
  Serum vascular endothelial growth factor levels in fasting were collected and measured.
procalcitonin | From enrollment to the end of treatment at 3rd month
  Serum procalcitonin levels in fasting were collected and measured.
Systemic Vascular Resistance | From enrollment to the end of treatment at 3rd month
  Stroke Systemic Vascular Resistance Index was collected and measured.
Mean Arterial Pressure | From enrollment to the end of treatment at 3rd month
  Mean Arterial Pressure was collected and measured.
Stroke Volume Index | From enrollment to the end of treatment at 3rd month
  Stroke Volume Index was collected and measured.
Stroke Volume | From enrollment to the end of treatment at 3rd month
  Stroke Volume levels was collected and measured.
Cardiac Output | From enrollment to the end of treatment at 3rd month
  Cardiac Output was collected and measured.
Cardiac Index | From enrollment to the end of treatment at 3rd month
  The Cardiac Index was collected and measured.
Left Ventricular Stroke Work Index | From enrollment to the end of treatment at 3rd month
  The left Ventricular Stroke Work Index was collected and measured.
Systemic Vascular Resistance Index | From enrollment to the end of treatment at 3rd month
  The systemic Vascular Resistance Index was collected and measured.
Ejection Phase Contraction Index | From enrollment to the end of treatment at 3rd month
  Ejection Phase Contraction Index was collected and measured.
Inotropic State Index | From enrollment to the end of treatment at 3rd month
  Inotropic State Index was collected and measured.
Systemic Vascular Resistance | From enrollment to the end of treatment at 3rd month
  Systemic Vascular Resistance was collected and measured.
Vascular Resistance | From enrollment to the end of treatment at 3rd month
  Vascular Resistance was collected and measured.
Mean Heart Rate | From enrollment to the end of treatment at 3rd month
  Mean Heart Rate was collected and measured.
left ventricular ejection fraction | From enrollment to the end of treatment at 3rd month
  left ventricular ejection fraction was collected and measured
Wall thickening fraction | From enrollment to the end of treatment at 3rd month
  Wall thickening fraction was collected and measured.
E/E' | From enrollment to the end of treatment at 3rd month
  E/E' was collected and measured.
6-minute walk test | From enrollment to the end of treatment at 3rd month
  A 6-minute walk test was collected and measured.
Patient Health Questionnaire-9 | From enrollment to the end of treatment at 3rd month
  Patient Health Questionnaire-9 was scored and collected. The Patient Health Questionnaire-9 (PHQ-9) serves as a critical instrument for the screening, diagnosis, and assessment of depression, enabling the measurement of its severity.
7-item Generalized Anxiety Disorder Scale | From enrollment to the end of treatment at 3rd month
  A 7-item Generalized Anxiety Disorder Scale (GAD-7) was scored and collected. GAD-7 acts as an essential tool for evaluating generalized anxiety disorder
The Pittsburgh Sleep Quality Index (PSQI) | From enrollment to the end of treatment at 3rd month
  The Pittsburgh Sleep Quality Index (PSQI)was scored and collected. the Pittsburgh Sleep Quality Index (PSQI) stands as a widely recognized assessment tool for determining sleep quality.
Seattle Angina Questionnaire (SAQ) | From enrollment to the end of treatment at 3rd month
  The Seattle Angina Questionnaire (SAQ) was scored and collected. SAQ functions as a self-administered assessment tool designed to evaluate specific functional status and quality of life among individuals with coronary artery disease.
Heart rate variability | From enrollment to the end of treatment at 3rd month
  Heart rate variability was scored and collected. Heart rate variability (HRV) refers to the fluctuation in the timing of consecutive heartbeats or the variance in heart rate. It is determined by the duration between two successive R-R intervals, representing the slight deviation between each cardiac cycle. HRV assessment was conducted using the ZSY-1 Rhythm Variability Analyzer, with the patient in a supine position, and short-term (5-minute) HRV was measured during daytime hours (8:00-16:00) while at rest.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Peng, MD, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinnan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
The study data is related to participant privacy. The data that support the findings of this study are available on request from the corresponding author [Lin Shen].

REFERENCES:
- [Result] Liang W, Liang B, Yan K, Zhang G, Zhuo J, Cai Y. Low-Intensity Pulsed Ultrasound: A Physical Stimulus with Immunomodulatory and Anti-inflammatory Potential. Ann Biomed Eng. 2024 Aug;52(8):1955-1981. doi: 10.1007/s10439-024-03523-y. Epub 2024 Apr 29. PMID 38683473
- [Result] Zhu H, He M, Wang YL, Zhang Y, Dong J, Chen BY, Li YL, Zhou LJ, Du LJ, Liu Y, Zhang WC, Ta D, Duan SZ. Low-intensity pulsed ultrasound alleviates doxorubicin-induced cardiotoxicity via inhibition of S100a8/a9-mediated cardiac recruitment of neutrophils. Bioeng Transl Med. 2023 Jul 7;8(6):e10570. doi: 10.1002/btm2.10570. eCollection 2023 Nov. PMID 38023700
- [Result] Watanabe T, Matsumoto Y, Nishimiya K, Shindo T, Amamizu H, Sugisawa J, Tsuchiya S, Sato K, Morosawa S, Ohyama K, Watanabe-Asaka T, Hayashi M, Kawai Y, Takahashi J, Yasuda S, Shimokawa H. Low-intensity pulsed ultrasound therapy suppresses coronary adventitial inflammatory changes and hyperconstricting responses after coronary stent implantation in pigs in vivo. PLoS One. 2021 Sep 13;16(9):e0257175. doi: 10.1371/journal.pone.0257175. eCollection 2021. PMID 34516572
- [Result] Signori LU, Rubin Neto LJ, Jaenisch RB, Puntel GO, Nunes GS, Paulitsch FS, Hauck M, Silva AMVD. Effects of therapeutic ultrasound on the endothelial function of patients with type 2 diabetes mellitus. Braz J Med Biol Res. 2023 Jun 26;56:e12576. doi: 10.1590/1414-431X2023e12576. eCollection 2023. PMID 37377306
- [Result] de Avila Santana L, Alves JM, Andrade TA, Kajiwara JK, Garcia SB, Gomes FG, Frade MA. Clinical and immunohistopathological aspects of venous ulcers treatment by Low-Intensity Pulsed Ultrasound (LIPUS). Ultrasonics. 2013 Apr;53(4):870-9. doi: 10.1016/j.ultras.2012.12.009. Epub 2012 Dec 23. PMID 23294989
- [Result] Shindo T, Ito K, Ogata T, Kurosawa R, Eguchi K, Kagaya Y, Hanawa K, Hasebe Y, Nishimiya K, Shiroto T, Takahashi J, Okumura Y, Noguchi T, Ozaki Y, Daida H, Hagiwara N, Masuyama T, Chikamori T, Fukumoto Y, Tsujita K, Kanai H, Yasuda S, Shimokawa H. A randomized, double-blind, placebo-controlled pilot trial of low-intensity pulsed ultrasound therapy for refractory angina pectoris. PLoS One. 2023 Jun 23;18(6):e0287714. doi: 10.1371/journal.pone.0287714. eCollection 2023. PMID 37352324
- [Result] Shindo T, Ito K, Ogata T, Hatanaka K, Kurosawa R, Eguchi K, Kagaya Y, Hanawa K, Aizawa K, Shiroto T, Kasukabe S, Miyata S, Taki H, Hasegawa H, Kanai H, Shimokawa H. Low-Intensity Pulsed Ultrasound Enhances Angiogenesis and Ameliorates Left Ventricular Dysfunction in a Mouse Model of Acute Myocardial Infarction. Arterioscler Thromb Vasc Biol. 2016 Jun;36(6):1220-9. doi: 10.1161/ATVBAHA.115.306477. Epub 2016 Apr 14. PMID 27079882
- [Result] Li J, Zhang Q, Ren C, Wu X, Zhang Y, Bai X, Lin Y, Li M, Fu J, Kopylov P, Wang S, Yu T, Wang N, Xu C, Zhang Y, Yang B. Low-Intensity Pulsed Ultrasound Prevents the Oxidative Stress Induced Endothelial-Mesenchymal Transition in Human Aortic Endothelial Cells. Cell Physiol Biochem. 2018;45(4):1350-1365. doi: 10.1159/000487561. Epub 2018 Feb 15. PMID 29462805
- [Result] Hu Y, Jia Y, Wang H, Cao Q, Yang Y, Zhou Y, Tan T, Huang X, Zhou Q. Low-intensity pulsed ultrasound promotes cell viability and inhibits apoptosis of H9C2 cardiomyocytes in 3D bioprinting scaffolds via PI3K-Akt and ERK1/2 pathways. J Biomater Appl. 2022 Sep;37(3):402-414. doi: 10.1177/08853282221102669. Epub 2022 May 15. PMID 35574901
- [Result] Sun P, Li Y, Yu W, Chen J, Wan P, Wang Z, Zhang M, Wang C, Fu S, Mang G, Choi S, Du Z, Tang C, Li S, Shi G, Tian J, Dai J, Leng X. Low-intensity pulsed ultrasound improves myocardial ischaemia-reperfusion injury via migrasome-mediated mitocytosis. Clin Transl Med. 2024 Jul;14(7):e1749. doi: 10.1002/ctm2.1749. PMID 38951127
- [Result] Weng L, Li L, Zhao K, Xu T, Mao Y, Shu H, Chen X, Chen J, Wu J, Guo X, Tu J, Zhang D, Sun W, Kong X. Non-Invasive Local Acoustic Therapy Ameliorates Diabetic Heart Fibrosis by Suppressing ACE-Mediated Oxidative Stress and Inflammation in Cardiac Fibroblasts. Cardiovasc Drugs Ther. 2022 Jun;36(3):413-424. doi: 10.1007/s10557-021-07297-6. Epub 2022 Feb 14. PMID 35156147
- [Result] Zhao K, Zhang J, Xu T, Yang C, Weng L, Wu T, Wu X, Miao J, Guo X, Tu J, Zhang D, Zhou B, Sun W, Kong X. Low-intensity pulsed ultrasound ameliorates angiotensin II-induced cardiac fibrosis by alleviating inflammation via a caveolin-1-dependent pathway. J Zhejiang Univ Sci B. 2021 Oct 15;22(10):818-838. doi: 10.1631/jzus.B2100130. PMID 34636186
- [Result] Zhao K, Weng L, Xu T, Yang C, Zhang J, Ni G, Guo X, Tu J, Zhang D, Sun W, Kong X. Low-intensity pulsed ultrasound prevents prolonged hypoxia-induced cardiac fibrosis through HIF-1alpha/DNMT3a pathway via a TRAAK-dependent manner. Clin Exp Pharmacol Physiol. 2021 Nov;48(11):1500-1514. doi: 10.1111/1440-1681.13562. Epub 2021 Aug 14. PMID 34343366
- [Result] Monma Y, Shindo T, Eguchi K, Kurosawa R, Kagaya Y, Ikumi Y, Ichijo S, Nakata T, Miyata S, Matsumoto A, Sato H, Miura M, Kanai H, Shimokawa H. Low-intensity pulsed ultrasound ameliorates cardiac diastolic dysfunction in mice: a possible novel therapy for heart failure with preserved left ventricular ejection fraction. Cardiovasc Res. 2021 Apr 23;117(5):1325-1338. doi: 10.1093/cvr/cvaa221. PMID 32683442
- [Result] Jiang X, Savchenko O, Li Y, Qi S, Yang T, Zhang W, Chen J. A Review of Low-Intensity Pulsed Ultrasound for Therapeutic Applications. IEEE Trans Biomed Eng. 2019 Oct;66(10):2704-2718. doi: 10.1109/TBME.2018.2889669. Epub 2018 Dec 25. PMID 30596564
- [Result] Cruz Rodriguez JB, Kar S. Management of Angina Post Percutaneous Coronary Intervention. Curr Cardiol Rep. 2020 Jan 21;22(2):7. doi: 10.1007/s11886-020-1259-9. PMID 31965355
- [Result] Tao S, Tang X, Yu L, Li L, Zhang G, Zhang L, Huang L, Wu J. Prognosis of coronary heart disease after percutaneous coronary intervention: a bibliometric analysis over the period 2004-2022. Eur J Med Res. 2023 Sep 1;28(1):311. doi: 10.1186/s40001-023-01220-5. PMID 37658418
- [Result] Ozaki Y, Tobe A, Onuma Y, Kobayashi Y, Amano T, Muramatsu T, Ishii H, Yamaji K, Kohsaka S, Ismail TF, Uemura S, Hikichi Y, Tsujita K, Ako J, Morino Y, Maekawa Y, Shinke T, Shite J, Igarashi Y, Nakagawa Y, Shiode N, Okamura A, Ogawa T, Shibata Y, Tsuji T, Hayashida K, Yajima J, Sugano T, Okura H, Okayama H, Kawaguchi K, Zen K, Takahashi S, Tamura T, Nakazato K, Yamaguchi J, Iida O, Ozaki R, Yoshimachi F, Ishihara M, Murohara T, Ueno T, Yokoi H, Nakamura M, Ikari Y, Serruys PW, Kozuma K; Task Force on Primary Percutaneous Coronary Intervention (PCI) of the Japanese Association of Cardiovascular Intervention, Therapeutics (CVIT). CVIT expert consensus document on primary percutaneous coronary intervention (PCI) for acute coronary syndromes (ACS) in 2024. Cardiovasc Interv Ther. 2024 Oct;39(4):335-375. doi: 10.1007/s12928-024-01036-y. Epub 2024 Sep 20. PMID 39302533
- [Result] Hoole SP, Bambrough P. Recent advances in percutaneous coronary intervention. Heart. 2020 Sep;106(18):1380-1386. doi: 10.1136/heartjnl-2019-315707. Epub 2020 Jun 10. PMID 32522821
- [Result] Roth GA, Mensah GA, Johnson CO, Addolorato G, Ammirati E, Baddour LM, Barengo NC, Beaton AZ, Benjamin EJ, Benziger CP, Bonny A, Brauer M, Brodmann M, Cahill TJ, Carapetis J, Catapano AL, Chugh SS, Cooper LT, Coresh J, Criqui M, DeCleene N, Eagle KA, Emmons-Bell S, Feigin VL, Fernandez-Sola J, Fowkes G, Gakidou E, Grundy SM, He FJ, Howard G, Hu F, Inker L, Karthikeyan G, Kassebaum N, Koroshetz W, Lavie C, Lloyd-Jones D, Lu HS, Mirijello A, Temesgen AM, Mokdad A, Moran AE, Muntner P, Narula J, Neal B, Ntsekhe M, Moraes de Oliveira G, Otto C, Owolabi M, Pratt M, Rajagopalan S, Reitsma M, Ribeiro ALP, Rigotti N, Rodgers A, Sable C, Shakil S, Sliwa-Hahnle K, Stark B, Sundstrom J, Timpel P, Tleyjeh IM, Valgimigli M, Vos T, Whelton PK, Yacoub M, Zuhlke L, Murray C, Fuster V; GBD-NHLBI-JACC Global Burden of Cardiovascular Diseases Writing Group. Global Burden of Cardiovascular Diseases and Risk Factors, 1990-2019: Update From the GBD 2019 Study. J Am Coll Cardiol. 2020 Dec 22;76(25):2982-3021. doi: 10.1016/j.jacc.2020.11.010. PMID 33309175
- [Result] Stone PH, Libby P, Boden WE. Fundamental Pathobiology of Coronary Atherosclerosis and Clinical Implications for Chronic Ischemic Heart Disease Management-The Plaque Hypothesis: A Narrative Review. JAMA Cardiol. 2023 Feb 1;8(2):192-201. doi: 10.1001/jamacardio.2022.3926. PMID 36515941
- [Derived] He C, Peng J, Liu H, Zhong L, Wei Y, Qiu H, Liu C, Lv N, Liu L, Qi X, Zhang F, You B, Song Q, Shen L. A study protocol of the rehabilitative efficacy of cardiovascular ultrasound therapy after percutaneous coronary intervention in patients with coronary artery disease: A multicenter, parallel-group, randomized controlled study. PLoS One. 2025 Oct 16;20(10):e0327557. doi: 10.1371/journal.pone.0327557. eCollection 2025. PMID 41100539